CLINICAL TRIAL: NCT04977817
Title: A Prospective/Retrospective Chart Review of the Effects of a Probiotic Dietary Supplement on Days of Total Parenteral Nutrition in Two Neonatal Intensive Care Units
Brief Title: Probiotics/TPN in the NICU
Status: Completed | Type: Observational
Sponsor: Pediatrix (Other)
Collaborators: Phoenix Children's Hospital (Other); Banner University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 822180615
Record Dates: First submitted 2021-06-28; First posted 2021-07-27 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Total Parenteral Nutrition; Necrotizing Enterocolitis of Newborn
MeSH Terms: conditions — Hyperphagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: By using the Baby Steps Program, neonates less than or equal to 1500 grams and less than 32 weeks GA will be identified. The control group will contain those that did not receive probiotics.
- Treatment Group: By using the Baby Steps Program, neonates less than or equal to 1500 grams and less than 32 weeks GA will be identified. The treatment group will contain those neonates that did receive the probiotic nutritional supplement.
  Interventions: Dietary Supplement: Similac Probiotic Tri-Blend

INTERVENTIONS:
Dietary Supplement: Similac Probiotic Tri-Blend — Probiotic dietary supplement, Similac Probiotic Tri-Blend
  Groups: Treatment Group

SUMMARY:
The purpose of this study is to evaluate the effect of probiotic administration on TPN dependence in infants < 32 weeks GA and BW 1500 grams or less in the Banner - University Medical Center Phoenix and Banner Children's at Desert Neonatal Intensive Care Units (NICU). The primary endpoint of capturing the number of days of TPN administration can reflect that an infant is progressing towards readiness for the initiation or advancement of enteral feedings at an earlier interval. The relationship between probiotic administration and the incidence of NEC, culture positive sepsis, and mortality is of interest to us and will be captured. Finally, the assessment of the tolerance of probiotic administration and the potential positive impact on growth and development in these premature infants may validate our current practices.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight < 1500 grams or GA < 32 weeks

Exclusion Criteria:

* Life threatening congenital anomalies
* Transfers to another facility prior to discharge home
* Investigator discretion to exclude if deemed necessary

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subject population will be infants admitted to the Banner - University Medical Center Phoenix and Banner Children's at Desert NICUs who meet the specific inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
Number of days on total parenteral nutrition | 30 days
  Evaluate the effects of a probiotic dietary supplement (Similac Probiotic Tri-Blend) on number of days on total parenteral nutrition (TPN) in infants admitted to the Neonatal Intensive Care Unit (NICU).

SECONDARY OUTCOMES:
Impact on neonatal growth | 30 days
  Neonatal growth velocity may be impacted by the usage of probiotics in the Neonatal Intensive Care Unit.
Feeding Intolerance | 30 days
  The administration of probiotics may change the incidence of feeding intolerance

OTHER OUTCOMES:
Incidence of NEC | 30 days
  Probiotic administration may change the incidence of Necrotizing Enterocolitis
Days on Respiratory Support | 30 days
  Days on respiratory support may represent an indication of overall outcomes in the Neonatal Intensive Care Unit
Incidence of culture positive sepsis | 30 days
  Probiotic administration may change the incidence of culture positive sepsis
Incidence of complication of central lines | 30 days
  Probiotic administration may change the length of time that a central line will need to be in place.
All causes of Mortality | 30 days
  Probiotic administration may change the incidence of mortality in the Neonatal Intensive Care Unit.

CONTACTS AND LOCATIONS:
Overall Officials: Suganya Kathiravan, MD, Principal Investigator — Phoenix Perinatal Associates - Neonatal Division
Locations (2):
- United States (2):
  - Banner Children's at Desert, Mesa, Arizona
  - Banner University Medical Center Phoenix, Phoenix, Arizona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jacobs SE, Tobin JM, Opie GF, Donath S, Tabrizi SN, Pirotta M, Morley CJ, Garland SM; ProPrems Study Group. Probiotic effects on late-onset sepsis in very preterm infants: a randomized controlled trial. Pediatrics. 2013 Dec;132(6):1055-62. doi: 10.1542/peds.2013-1339. Epub 2013 Nov 18. PMID 24249817
- [Background] Gray KD, Messina JA, Cortina C, Owens T, Fowler M, Foster M, Gbadegesin S, Clark RH, Benjamin DK Jr, Zimmerman KO, Greenberg RG. Probiotic Use and Safety in the Neonatal Intensive Care Unit: A Matched Cohort Study. J Pediatr. 2020 Jul;222:59-64.e1. doi: 10.1016/j.jpeds.2020.03.051. Epub 2020 May 14. PMID 32418818
- [Background] Patel RM, Underwood MA. Probiotics and necrotizing enterocolitis. Semin Pediatr Surg. 2018 Feb;27(1):39-46. doi: 10.1053/j.sempedsurg.2017.11.008. Epub 2017 Nov 6. PMID 29275816
- [Background] Singh B, Shah PS, Afifi J, Simpson CD, Mitra S, Dow K, El-Naggar W; Canadian Neonatal Network Investigators. Probiotics for preterm infants: A National Retrospective Cohort Study. J Perinatol. 2019 Apr;39(4):533-539. doi: 10.1038/s41372-019-0315-z. Epub 2019 Jan 28. PMID 30692619
- [Background] Sawh SC, Deshpande S, Jansen S, Reynaert CJ, Jones PM. Prevention of necrotizing enterocolitis with probiotics: a systematic review and meta-analysis. PeerJ. 2016 Oct 5;4:e2429. doi: 10.7717/peerj.2429. eCollection 2016. PMID 27761306